CLINICAL TRIAL: NCT01515917
Title: Citicoline and Omega-3 Fatty Acid Effects in Veterans With TBI
Brief Title: Citicoline and Omega-3 Fatty Acid Effects in Veterans With Traumatic Brain Injury (TBI)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Yurgelun-Todd (Other)
Responsible Party: Sponsor-Investigator, Deborah Yurgelun-Todd, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_53174
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Traumatic Brain Injury; Substance Abuse; Substance Dependence
Keywords: Veterans; Traumatic Brain Injury; TBI; Substance Abuse; Substance Dependence; Veterans with traumatic brain injury (TBI); Veterans with substance abuse or dependence
MeSH Terms: conditions — Brain Injuries, Traumatic; Substance-Related Disorders | interventions — Cytidine Diphosphate Choline; Docosahexaenoic Acids; Rice Bran Oil; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citicoline and Omega-3 (Experimental): At visit 1 and again at visit 2, participants assigned to the experimental arm will receive a 14-day supply of citicoline and omega-3 fatty acid, of which they will be instructed to take 1000 mg and 2000 mg daily, respectively. This will be done in a double-blind, randomized fashion.
  Interventions: Drug: Citicoline; Drug: Omega-3
- Placebo (Placebo Comparator): At visit 1 and again at visit 2, participants assigned to the placebo group will be given 14-day supplies of placebo to be taken daily throughout the study period. This will be done in a double-blind, randomized fashion.
  Interventions: Other: Rice bran oil; Other: Microcrystalline Cellulose

INTERVENTIONS:
Drug: Citicoline — Participants randomly assigned to the experimental group, who, in addition to the research staff will be blind to such assignment, will be instructed to orally administer 1000 mg daily citicoline. These participants will receive a 14-day supply of citicoline at visit 1 and again at visit 2, making for a 28-day administration period.
  Other Names: Cognizin Citicoline
  Arms: Citicoline and Omega-3
Drug: Omega-3 — Participants randomly assigned to the experimental group, who, in addition to the research staff will be blind to such assignment, will be instructed to orally administer 2000 mg daily omega-3. These participants will receive a 14-day supply of omega-3 at visit 1 and again at visit 2, making for a 28-day administration period.
  Other Names: Omegabrite
  Arms: Citicoline and Omega-3
Other: Rice bran oil — Rice bran oil will be one of two placebos administered to participants randomly assigned to the placebo arm. Rice bran oil will serve as the placebo for omega-3 fatty acids and will be orally administered daily in 500 mg doses.
  Arms: Placebo
Other: Microcrystalline Cellulose — Microcrystalline Cellulose will be one of two placebos administered to participants randomly assigned to the placebo arm. Microcrystalline Cellulose will serve as the placebo for Citicoline and will be orally administered daily in 470 mg doses.
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study intended to examine the effects of the neutraceutical citicholine, together with omega-3 fatty acids, on a range of measures in individuals with concussive head injury, often referred to as traumatic brain injury, or TBI. The study will consist of three visits, during which participants will complete brain scans, a thorough testing battery and a clinical interview to assess mood and other diagnostic information relevant to the study.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Age 18 to 55
* History of TBI
* DSM-IV-TR diagnosis of abuse or dependence disorder for either alcohol or drugs of abuse
* Multiple concussive head injuries that meet the following criteria for TBI: 1) normal structural imaging, 2) loss of consciousness (LOC) between 0-30 minutes, 3) alteration of consciousness or mental status for a moment up to 2 hours or 4) post-traumatic amnesia of 0-1 day
* Stable on current psychotropic medication regimen for ≥ 3 months

Exclusion Criteria:

* Non Veteran
* Significant medical or neurological illness with the exception of TBI, which might affect cognitive function
* Significant medical illness which has the potential to be exacerbated by ingestion of citicoline/omega-3 fatty acids, including diabetes, congestive heart disorder, hyperlipidemia and severe coronary artery disease
* Age other than 18 to 55 years old
* History of ECT treatment
* Estimated IQ < 70
* Past or present history of bipolar disorder, schizophrenia, delusional disorder or any other psychotic disorder
* Currently taking a prescribed blood thinner (i.e., Coumadin)
* Claustrophobia
* Metal implanted within the body
* Pregnancy or lactation
* Left-handedness
* Poor vision, as subjects must have normal or corrected-to-normal vision for viewing of cognitive challenge paradigms during fMRI protocols
* Non-native English speakers (for neurocognitive tasks)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive performance | 28 days
  Using baseline assessment measures gathered at Visit 1, assessments collected at Visits 2 and 3 will be used to determine whether the combined administration of neutraceuticals citicoline and omega-3 fatty acids will improve neurocognitive performance in individuals with TBI and substance abuse/dependence.

SECONDARY OUTCOMES:
Brain changes | 28 days
  Participants will undergo MRI scanning designed to assess white matter microstructure and focal brain activation at Visit 1 (Day 0) and again at Visit 3 (Day 28) in order to determine whether the combined administration of neutraceuticals citicoline and omega-3 fatty acids result in changes to these brain indices in participants with TBI and substance abuse/dependence.